CLINICAL TRIAL: NCT04710966
Title: Comparison Between Arthroscopic Debridement and Repair for Ellman Grade II Bursal-side Partial-thickness Rotator Cuff Tears: a Prospective Randomized Controlled Trial
Brief Title: Comparison Between Arthroscopic Debridement and Repair for Partial-thickness Rotator Cuff Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: wangteng
Record Dates: First submitted 2021-01-06; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Rotator Cuff Tears
Keywords: partial-thickness; bursal-side tear; rotator cuff tears; arthroscopic debridement; arthroscopic repair
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Before initiating the trial, an investigator who was not involved in the study generated a computer-generated randomization list (block length 10, ratio 1:1). Allocation concealment was achieved by using opaque, sealed, sequentially numbered envelopes containing details of group assignment. Assignment occurred after baseline information was recorded. According to preoperative allocation, the patients were given arthroscopic debridement or repair respectively.For the debridement group, only stump refreshing and surrounding soft tissue cleaning were performed. For the repair group, we converted partial tears into full-thickness tears and sutured them
Who Masked: Outcomes Assessor
Masking Description: Whereas patients and surgeons were aware of the group assignments, the outcome assessors and data analysts were remained blinded during the study period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- debridement group (Experimental): For the debridement group, if the tear type is confirmed to be bursal-side Ellman grade II during the operation, arthroscopic debridement will be performed.
  Interventions: Procedure: arthroscopic debridement
- repair group (Experimental): For the repair group, if the tear type is confirmed to be bursal-side Ellman grade II during the operation, arthroscopic repair will be performed.
  Interventions: Procedure: arthroscopic repair

INTERVENTIONS:
Procedure: arthroscopic debridement — For the arthroscopic debridement, only stump refreshing and surrounding soft tissue cleaning were performed.
  Arms: debridement group
Procedure: arthroscopic repair — For the arthroscopic repair, we converted partial tears into full-thickness tears and sutured them.
  Arms: repair group

SUMMARY:
The purpose of this study is to conduct a prospective randomized controlled trial to compare the effects of arthroscopic debridement and repair for Ellman grade II bursal-side partial-thickness rotator cuff tears.The hypothesis was that there would be no difference in prognosis between arthroscopic debridement and repair.

DETAILED DESCRIPTION:
This was a single-center, prospective, double-blinded, randomized controlled trial, comparing arthroscopic debridement and arthroscopic repair for Ellman grade II BPTRCTs. Participants were recruited from September 2017 to April 2019. Before initiating the trial, an investigator who was not involved in the study generated a computer-generated randomization list (block length 10, ratio 1:1). Allocation concealment was achieved by using opaque, sealed, sequentially numbered envelopes containing details of group assignment. Assignment occurred after baseline information was recorded. Whereas participants and surgeons were aware of the group assignments, the outcome assessors and data analysts were remained blinded during the study period. Operations were performed by the same team of sports medicine surgeons under general anesthesia. For the debridement group, only stump refreshing and surrounding soft tissue cleaning were performed. For the repair group, partial tears were converted into full-thickness tears and sutured. The sample size calculation was based on data from previous studies, where the difference in Constant-Murray Shoulder (CMS) score between patients with arthroscopic repair and arthroscopic debridement was 8.81 points (93.90 vs. 85.09) with standard deviations of 5.4 and 21. Accepting an α risk of 0.05 and a β risk of 0.2 in a bilateral contrast, the minimum sample size required for each group was 35. To compensate for an estimated 15% loss to follow up, at least 82 patients would be included.

ELIGIBILITY:
Inclusion Criteria:

* Bursal-side partial-thickness rotator cuff tears (BPTRCTs) revealed by magnetic resonance imaging (MRI)
* Failed of conservative treatment for more than 3 months
* Intraoperative arthroscopic confirmed that the tear was Ellman grade II

Exclusion Criteria:

* Previous surgical surgery on the shoulder
* Articular-side or intratendinous rotator cuff tears
* Combined articular-side partial-thickness rotator cuff tears(APRCTs) and Bursal-side partial-thickness rotator cuff tears (BPRCTs), or full-thickness rotator cuff tears (RCTs)
* Combined with other shoulder lesions that need to be addressed, such as biceps tendon disorders, labral tears
* The presence of other diseases that affect shoulder function
* Contraindication to arthroscopic surgery or anesthesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
The Visual Analog Scale score | Baseline
  Assess pain on a scale of 0 (no pain) to 10 (worst possible pain).
The Visual Analog Scale score | Postoperative 6 months
  Assess pain on a scale of 0 (no pain) to 10 (worst possible pain).
The Visual Analog Scale score | Postoperative 12 months
  Assess pain on a scale of 0 (no pain) to 10 (worst possible pain).
The Visual Analog Scale score | Postoperative 18 months
  Assess pain on a scale of 0 (no pain) to 10 (worst possible pain).
Constant-Murray Shoulder score | Baseline
  An assessment method often used by orthopedic surgeons when assessing the condition of patients with shoulder joints. Possible scores range from 0 to 100，a higher score means a better result.
Constant-Murray Shoulder score | postoperative 6 months
  An assessment method often used by orthopedic surgeons when assessing the condition of patients with shoulder joints.Possible scores range from 0 to 100，a higher score means a better result.
Constant-Murray Shoulder score | postoperative 12 months
  An assessment method often used by orthopedic surgeons when assessing the condition of patients with shoulder joints.Possible scores range from 0 to 100，a higher score means a better result.
Constant-Murray Shoulder score | postoperative 18 months
  An assessment method often used by orthopedic surgeons when assessing the condition of patients with shoulder joints.Possible scores range from 0 to 100，a higher score means a better result.
American Shoulder and Elbow Surgeon score | Baseline
  The evaluation criteria used to assess shoulder joint function based on the patients' pain and accumulated daily activities. Possible scores range from 0 to 100. The higher the score, the better the shoulder joint function.
American Shoulder and Elbow Surgeon score | postoperative 6 months
  The evaluation criteria used to assess shoulder joint function based on the patients' pain and accumulated daily activities. Possible scores range from 0 to 100. The higher the score, the better the shoulder joint function.
American Shoulder and Elbow Surgeon score | postoperative 12 months
  The evaluation criteria used to assess shoulder joint function based on the patients' pain and accumulated daily activities. Possible scores range from 0 to 100. The higher the score, the better the shoulder joint function.
American Shoulder and Elbow Surgeon score | postoperative 18 months
  The evaluation criteria used to assess shoulder joint function based on the patients' pain and accumulated daily activities. Possible scores range from 0 to 100. The higher the score, the better the shoulder joint function.
University of California-Los Angeles score | Baseline
  The score mainly consists of two parts. Patients subjectively evaluate pain and functional activity; and doctors objectively evaluate shoulder joint mobility and muscle strength. Possible scores range from 0 to 35, a higher score means a better result.
University of California-Los Angeles score | postoperative 6 months
  The score mainly consists of two parts. Patients subjectively evaluate pain and functional activity; and doctors objectively evaluate shoulder joint mobility and muscle strength. Possible scores range from 0 to 35, a higher score means a better result.
University of California-Los Angeles score | postoperative 12 months
  The score mainly consists of two parts. Patients subjectively evaluate pain and functional activity; and doctors objectively evaluate shoulder joint mobility and muscle strength. Possible scores range from 0 to 35, a higher score means a better result.
University of California-Los Angeles score | postoperative 18 months
  The score mainly consists of two parts. Patients subjectively evaluate pain and functional activity; and doctors objectively evaluate shoulder joint mobility and muscle strength. Possible scores range from 0 to 35, a higher score means a better result.

SECONDARY OUTCOMES:
Grading of rotator cuff integrity | 18 months after surgery
  The integrity of the rotator cuff was assessed by magnetic resonance imaging (MRI) according to a grading criteria, as follows: Grade I and II, sufficient thickness with low or partial high intensity; Grade III, insufficient thickness without discontinuity; Grade IV and V, presence of a minor or major discontinuity.
Grading of muscle atrophy | 18 months after surgery
  Muscular atrophy was assessed on oblique sagittal MRI images using an occupation ratio measured by dividing the supraspinatus muscle's cross-sectional area by that of the supraspinatus fossa on the oblique-sagittal view. When the ratio was between 1.00 and 0.60, the muscle was considered normal or with slight atrophy (Grade I); values between 0.60 and 0.40 indicated moderate atrophy (Grade II); values below 0.40 indicated severe atrophy (Grade III).
Grading of fatty degeneration | 18 months after surgery
  Fatty degeneration in supraspinatus muscle was assessed by magnetic resonance imaging (MRI) according to a grading system with stages 0-4 as follows: grade 0, no fat; Grade 1, thin fatty streaks; Grade 2, heavy fat infiltration, with muscle still pre-dominating; Grade 3, even distribution of fat and muscle; Grade 4, more fat than muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Teng Wang, Principal Investigator — Investigator; Tengbo Yu, Study Chair — professor
Locations (1):
- Affiliated Hospital of Qingdao University, Qingdao, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Proposals should be directed to wt10113277@163.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website .
URL: http://www.medresman.org.cn/uc/sindex.aspx

REFERENCES:
- [Result] Ellman H. Diagnosis and treatment of incomplete rotator cuff tears. Clin Orthop Relat Res. 1990 May;(254):64-74. PMID 2182260
- [Result] Chung SW, Kim JY, Yoon JP, Lyu SH, Rhee SM, Oh SB. Arthroscopic repair of partial-thickness and small full-thickness rotator cuff tears: tendon quality as a prognostic factor for repair integrity. Am J Sports Med. 2015 Mar;43(3):588-96. doi: 10.1177/0363546514561004. Epub 2014 Dec 22. PMID 25535097
- [Result] Kwon OS, Kelly JI. Outcome analysis of arthroscopic treatment of partial thickness rotator cuff tears. Indian J Orthop. 2014 Jul;48(4):385-9. doi: 10.4103/0019-5413.136249. PMID 25143642
- [Result] Strauss EJ, Salata MJ, Kercher J, Barker JU, McGill K, Bach BR Jr, Romeo AA, Verma NN. Multimedia article. The arthroscopic management of partial-thickness rotator cuff tears: a systematic review of the literature. Arthroscopy. 2011 Apr;27(4):568-80. doi: 10.1016/j.arthro.2010.09.019. PMID 21296545
- [Result] Cordasco FA, Backer M, Craig EV, Klein D, Warren RF. The partial-thickness rotator cuff tear: is acromioplasty without repair sufficient? Am J Sports Med. 2002 Mar-Apr;30(2):257-60. doi: 10.1177/03635465020300021801. PMID 11912097
- [Result] Wolff AB, Magit DP, Miller SR, Wyman J, Sethi PM. Arthroscopic fixation of bursal-sided rotator cuff tears. Arthroscopy. 2006 Nov;22(11):1247.e1-4. doi: 10.1016/j.arthro.2006.05.026. PMID 17084305
- [Result] Zhang Y, Zhai S, Qi C, Chen J, Li H, Zhao X, Yu T. A comparative study of arthroscopic debridement versus repair for Ellman grade II bursal-side partial-thickness rotator cuff tears. J Shoulder Elbow Surg. 2020 Oct;29(10):2072-2079. doi: 10.1016/j.jse.2020.03.006. Epub 2020 Jun 1. PMID 32499197